CLINICAL TRIAL: NCT06521944
Title: CorEvitas RSV Vaccine Pregnancy Registry (RSV-PR)
Brief Title: RSV Vaccine Pregnancy Registry
Acronym: RSV-PR
Status: Recruiting | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: PRSV-300
Record Dates: First submitted 2024-07-16; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: Pregnant; Registry; RSV; RSV Vaccine; Respiratory Syncytial Virus; Infections; Virus Diseases; Lung Diseases; Respiratory Tract Diseases
MeSH Terms: conditions — Infections; Virus Diseases; Lung Diseases; Respiratory Tract Diseases | interventions — Respiratory Syncytial Virus Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed: Participants who receive RSV vaccine between 32 weeks, 0 days and 36 weeks, 6 days of gestation
  Interventions: Biological: RSV Vaccine
- Unexposed: Participants who do not receive RSV vaccine during pregnancy
  Interventions: Other: Non-exposure to RSV Vaccine

INTERVENTIONS:
Biological: RSV Vaccine — RSV Vaccine approved for administration to pregnant individuals between 32 weeks, 0 days and 36 weeks, 6 days of gestation
  Groups: Exposed
Other: Non-exposure to RSV Vaccine — Pregnant individuals who are not exposed to the RSV vaccine
  Groups: Unexposed

SUMMARY:
The research question is: What is the risk of adverse pregnancy outcomes, including preterm birth, hypertensive disorders, and other maternal and neonatal/infant outcomes, following exposure to RSV vaccine between 32 weeks, 0 days and 36 weeks, 6 days of gestation in the CorEvitas Respiratory Syncytial Virus Vaccine Pregnancy Registry (RSV-PR)? The primary study objective is to estimate the risk of (1) preterm birth and (2) hypertensive disorders following exposure to RSV vaccine between 32 weeks, 0 days and 36 weeks, 6 days of gestation.

The secondary study objective is to estimate the risk of other safety outcomes of interest following exposure to RSV vaccine between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including:

* Pregnancy-related outcomes: stillbirth, premature labor, premature rupture of membranes, preterm premature rupture of membranes, cesarean delivery, prolonged maternal duration of hospital stay
* Maternal outcomes: thrombocytopenia, Guillain-Barré syndrome, other immune-mediated demyelinating conditions, polyneuropathies, atrial fibrillation, maternal death
* Neonatal/infant outcomes: small for gestational age, large for gestational age, low birth weight, admission to a neonatal intensive care unit (NICU), NICU duration of stay, mechanical ventilation in neonatal period, neonatal death, postnatal growth at 1 year of age The exploratory study objective is to describe the most frequently reported maternal adverse events following exposure to RSV vaccine between 32 weeks, 0 days and 36 weeks, 6 days of gestation.

DETAILED DESCRIPTION:
Rationale and background: Respiratory syncytial virus (RSV) vaccine is approved for use in pregnant individuals during late pregnancy (32 weeks, 0 days through 36 weeks, 6 days of gestation) to prevent RSV-related severe lower respiratory tract disease in infants from birth through 6 months of age.

Research question and objectives: This work is intended to answer the question regarding what is the risk of adverse pregnancy outcomes, including preterm birth, hypertensive disorders, and other maternal and neonatal/infant outcomes, following exposure to RSV vaccine between 32 weeks, 0 days and 36 weeks, 6 days of gestation? The primary study objective is to estimate the risk of (1) preterm birth and (2) hypertensive disorders of pregnancy following exposure to RSV vaccine between 32 weeks, 0 days and 36 weeks, 6 days of gestation.

The secondary study objective is to estimate the risk of other safety outcomes of interest following exposure to RSV vaccine between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including:

* Pregnancy-related outcomes: stillbirth, premature labor, premature rupture of membranes (PROM), preterm premature rupture of membranes (PPROM), cesarean delivery, prolonged maternal duration of hospital stay
* Maternal outcomes: thrombocytopenia, Guillain-Barré syndrome (GBS), other immune-mediated demyelinating conditions, polyneuropathies, atrial fibrillation, maternal death
* Neonatal/infant outcomes: small for gestational age (SGA), large for gestational age, low birth weight (LBW), admission to a neonatal intensive care unit (NICU), NICU duration of stay, mechanical ventilation in neonatal period, neonatal death, postnatal growth deficiency at 1 year of age The exploratory study objective is to describe the most frequently reported maternal adverse events (AEs) occurring within 42 days of RSV vaccine administration between 32 weeks, 0 days and 36 weeks, 6 days of gestation.

Outcomes occurring before 32 weeks, 0 days of gestation, including but not limited to spontaneous abortion and major congenital malformations, will not be evaluated.

Study design: This US-based observational cohort study is designed to evaluate RSV vaccine exposure during weeks 32 through 36 of pregnancy (i.e., 32 weeks, 0 days through 36 weeks, 6 days) and the risk of subsequent pregnancy, maternal, and neonatal/infant outcomes. For this study, the index date will be the date of RSV vaccine administration for the exposed cohort and the date of enrollment for the unexposed cohort. The risks of pregnancy-related outcomes, maternal outcomes, and neonatal/infant outcomes for participants exposed and unexposed to RSV vaccine during pregnancy will be estimated.

Population: The study population will include 2 cohorts of individuals enrolled in the Respiratory Syncytial Virus Vaccine Pregnancy Registry (RSV-PR): (1) those exposed to RSV vaccine between 32 weeks, 0 days and 36 weeks, 6 days and (2) those unexposed to RSV vaccine during pregnancy.

Variables: Exposure to RSV vaccine will be defined as receipt of RSV vaccine at any time between 32 weeks, 0 days and 36 weeks, 6 days of gestation. The primary outcomes are preterm birth and hypertensive disorders of pregnancy. Secondary pregnancy outcomes of interest include stillbirth, premature labor, PROM, PPROM, cesarean delivery, and prolonged maternal duration of hospital stay. Maternal outcomes of interest include thrombocytopenia, GBS, other immune-mediated demyelinating conditions, polyneuropathies, atrial fibrillation, and maternal death. The neonatal/infant outcomes of interest are SGA, large for gestational age, LBW, admission to a NICU, prolonged infant duration of hospital stay, mechanical ventilation in neonatal period, neonatal death, and postnatal growth deficiency at 1 year of age. Maternal AEs occurring within 42 days of RSV vaccine administration will be captured for the cohort of RSV vaccine-exposed pregnant individuals.

Information on covariates (including demographics, risk factors for the study outcomes, comorbidities, concomitant medications, and predictors of RSV vaccine use) will be incorporated into the analyses.

Data source: This study will collect data from participants and the healthcare providers (HCPs) involved in their care or the care of their infants via concise data collection forms at pre-defined timepoints during pregnancy, at pregnancy outcome, and up to 1 year of infant age.

Study Size: The study will aim to include 2,062total participants (1,031 per cohort) to detect a minimum risk ratio of 1.5 or greater for the primary outcome of preterm birth (fewer participants are required to detect hypertensive disorders of pregnancy), assuming equal accrual (1:1) of RSV vaccine-exposed and -unexposed participants, and accounting for exclusions from the analysis population and loss of effective sample size due to inverse probability of treatment weighting.

Data analysis: Participant characteristics will be summarized with descriptive statistics for each cohort. Comparative analyses will be conducted for each outcome if sample size permits. Supplementary analyses will be conducted that include pregnant individuals who were excluded from the analysis population (i.e., those lacking HCP confirmation of RSV vaccine exposure, pregnancy, or outcomes of interest). If sample size permits, subgroup and sensitivity analyses will be performed to examine the extent to which changes in certain methods or assumptions affect the results.

Milestones: Start of data collection is planned for 30 September 2024, and the end of data collection is planned for 30 September 2030. The final study report and analysis is projected for 30 September 2031.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet the following inclusion criteria to be eligible for inclusion in the study:

  1. A resident of the US at enrollment
  2. 18 to 50 years of age at enrollment
  3. Gestational age of ≥32 weeks, 0 days at enrollment
  4. If exposed to RSV vaccine, receipt of any RSV vaccine between 32 weeks, 0 days and 36 weeks, 6 days of gestation
  5. Evidence of a personally signed and dated informed consent document or, upon waiver of written consent by the relevant IRB/independent ethics committee, verbal consent indicating that the individual (or a legally acceptable representative) has been informed of all pertinent aspects of the study
  6. Authorization obtained for the relevant HCP(s) to provide data to the registry
  7. Contact information available (for participant and HCPs)

Exclusion Criteria:

* Individuals meeting any of the following criteria will not be included in the study:

  1. Receipt of an RSV vaccine during pregnancy before 32 weeks, 0 days gestation
  2. Multi-fetal pregnancy
  3. Enrolled in the RSV-PR with a previous pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant individuals across the US who learn of the study via a nationwide advertising campaign or via their health care providers or maternal care sites
Sampling Method: Non-Probability Sample
Enrollment: 2062 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Risk of preterm birth following RSV vaccine exposure | 36 weeks, 6 days
  Risk of preterm birth following exposure to RSV vaccine between 32 weeks, 0 days and 36 weeks, 6 days of gestation
Risk of hypertensive disorders following RSV vaccine exposure | 42 days after date of vaccination
  Risk of hypertensive disorders following exposure to RSV vaccine between 32 weeks, 0 days and 36 weeks, 6 days of gestation

SECONDARY OUTCOMES:
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Pregnancy-related outcome: stillbirth
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Pregnancy-related outcome: premature labour
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Pregnancy-related outcome: premature rupture of membranes
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Pregnancy-related outcome: preterm premature rupture of membranes
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Pregnancy-related outcome: cesarean delivery
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Pregnancy-related outcome: prolonged maternal duration of hospital stay
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Maternal outcome: thrombocytopenia
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Maternal outcome: Guillain-Barré syndrome
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Maternal outcome: other immune-mediated demyelinating conditions
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Maternal outcome: polyneuropathies
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Maternal outcome: atrial fibrillation
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Maternal outcome: maternal death
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Neonatal/infant outcome: small for gestational age
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Neonatal/infant outcome: large for gestational age
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Neonatal/infant outcome: low birth weight
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Neonatal/infant outcome: admission to a neonatal intensive care unit (NICU)
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Neonatal/infant outcome: neonatal intensive care unit (NICU) duration of stay
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Neonatal/infant outcome: mechanical ventilation in neonatal period
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Neonatal/infant outcome: neonatal death
Risk of other safety outcomes of interest following RSV vaccine exposure | 42 days after date of vaccination
  The risk of other safety outcomes of interest following exposure to RSV vaccine as per routine clinical practice between 32 weeks, 0 days and 36 weeks, 6 days of gestation, including Neonatal/infant outcome: postnatal growth at 1 year of age
Frequently reported maternal adverse events following RSV vaccine exposure | 42 days after date of vaccination
  The most frequently reported maternal adverse events following exposure to RSV vaccine between 32 weeks, 0 days and 36 weeks, 6 days of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Ronna Chan, PhD, MPH, Principal Investigator — PPD, Part of Thermo Fisher Scientific
Locations (1):
- PPD, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://RSVPregnancyRegistry.com